CLINICAL TRIAL: NCT06355726
Title: Efficacy of Plasma Exchange Therapy vs Standard Medical Therapy in Severe Alcoholic Hepatitis With High Discriminant Function : A Randomised Controlled Trial
Brief Title: Efficacy of Plasma Exchange Therapy vs Standard Medical Therapy in Severe Alcoholic Hepatitis With High Discriminant Function
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Alcoholic Hepatitis-03
Record Dates: First submitted 2024-03-04; First posted 2024-04-09 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-02

CONDITIONS: Alcoholic Hepatitis
MeSH Terms: conditions — Hepatitis, Alcoholic | interventions — Plasma Exchange

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PLEX with SMT (Experimental): 3 sessions to 5 max, alternate day with SMT
  Interventions: Biological: Plasma Exchange; Other: Standard Medical Treatment
- SMT (Active Comparator): High calorie intake 35 to 40 Kcal/kg, protein 1.2 to 1.5 g/kg,albumin,antibiotics as required
  Interventions: Other: Standard Medical Treatment

INTERVENTIONS:
Biological: Plasma Exchange — Plasma exchange session will be done on alternate day to a maximum of 5 sessions. PLEX will be discontinued if the patients Shows sustained clinical improvement, Receive liver transplantation, Refuses further PLEX session,no improvement in clinical condition and Intolerant to PLEX procedure
  Arms: PLEX with SMT
Other: Standard Medical Treatment — Standard Medical Treatment

SUMMARY:
Alcoholic hepatitis, the most florid form of alcoholic liver disease, has a very high short-term mortality of up to 50% and no specific therapies are available other than steroids. Steroids also only show a limited utility in improving the short-term survival and boast no evidence of any long-term benefits. Additionally, only a small proportion of patients with alcoholic hepatitis are eligible to receive steroids. Thus, a large number of patients are either not eligible or do not respond to steroids and this group outnumbers those who do respond to steroids, leaving us without any specific therapeutic options for a majority of these individuals.[1] Even liver transplantation is not feasible in most cases due to the presence of sepsis or recent alcohol consumption and many ethical and logistic issues are involved despite the documented safety and survival benefits of early liver transplantation in patients with severe alcoholic hepatitis (SAH) not responding to medical management.[2,8] Therefore, newer, more effective, and nontransplant therapeutic options for managing severe alcoholic hepatitis are needed. TPE is expected to be an effective and well-tolerated bridge therapy in patients with severe alcoholic hepatitis of moderate severity not improving on SMT and without immediate prospects for liver transplantation.

DETAILED DESCRIPTION:
Hypothesis:wehypothesise that the early treatment with therapeutic plasma exchange in alcoholic hepatitis patients might improve overall survival in carefully selected patients by removing cytokines, chemokines and toxic substances.

Aim:

To compare transplant free survival between plasma exchange therapy and standard medical therapy in severe alcoholic hepatitis

Methodology:

Severe alcoholic hepatitis will be screened for the study and will be managed with SMT initially will be assessed for steroid therapy if becomes ineligible counselled for liver transplant in view of high DF and MELD ,if there is no options of Liver transplant in near future ,1 month will be given option for PLEX but it will be decided by randomisation whether he will get SMT or PLEX.He/she will also be told that PLEX is not a approved treatment and is a trial therapy and they may or may not get benefited.Patients Patients who agreed to undergo PLEX then undergo randomisation between PLEX and SMT and allocated in either group accordingly.

Control group will be administered SMT only.Case are those who get both SMT and PLEX. SMT involved empirical antibiotics as per treating physician,multivitamins,albumin. Hepatic encephalopathy (HE) will be treated with lactulose and rifaximin. Ascites with diuretics if not contraindicated because of renal insufficiency or HE. All patients will receive salt restricted, high protein diet (1.5 g/kg of proteins) either enterally/parenterally in addition to thiamine and multivitamins,35 to 45 kcal /kg .

Cases will be administered SMT with Plasma exchange session which will be done on alternate day to a maximum of 5 sessions. PLEX will be discontinued if the patients Shows sustained clinical improvement, Receive liver transplantation, Refuses further PLEX session,no improvement in clinical condition and Intolerant to PLEX procedure

Study population:

* Age - 18-60 years
* Patients with steroid ineligible(DF > 80< 120,MELD > 30) severe alcoholic hepatitis(Bili > 5 ,INR > 1.5)

Study design: Randomised controlled study done at Department of Hepatology,Institute of Liver and Biliary Sciences,NewDelhi,India.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 60 years
2. Severe alcoholic hepatitis with DF>80< 120 or MELD >30
3. No liver transplant option available in near future(for atleast 1 month)
4. Patient able to bear the cost of Plasma exchange by himself/herself

Exclusion Criteria:

1. Active sepsis
2. S creatinine >1.5mg/dl
3. Chronic kidney disease
4. Pregnancy
5. HCC or any other malignancy
6. Active Bleeding
7. Allergic to replacement fluid (FFP) in TPE
8. Severe Hypocalcemia (<7.6 mg/dl)
9. Failure to give consent
10. Financial issues to bear cost of Plasma exchange

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-09 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Liver transplant free survival at 28 days, 90 days and 180 days. | 28 days, 90 days and 180 days

SECONDARY OUTCOMES:
Change in total bilirubin and INR as measured by Discriminant Functions | 28 days, 90 days and 180 days
Number of patients with change in Model for End Stage Liver Disease (MELD) | 28 days, 90 days and 180 days
Number of patients with change in CTP | 28 days, 90 days and 180 days
Number of patients with change in LSM,SSM | 28 days, 90 days and 180 days
Mortality in both groups | 28 days, 90 days and 180 days
clinical improvement in the form of jaundice as measured by total bilirubin | 28 days, 90 days and 180 days
clinical improvement in the form of hepatic encephalopathy as measured by west haven criteria | 28 days, 90 days and 180 days
clinical improvement in the form of ascites as measured by ICA criteria. | 28 days, 90 days and 180 days
Frequency of decompensation events on follow up period | 28 days, 90 days and 180 days
Adverse events during plasma exchange | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences (ILBS), New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided